CLINICAL TRIAL: NCT06049407
Title: Intervention Through an Intelligent Technological Platform for Social-emotional Development and the Promotion of Well-being in Adolescence and Early Adulthood
Brief Title: Intervention on Socio-emotional Development and Well-being Through ICTs in Early Adulthood
Acronym: EMOWELL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Inmaculada Montoya Castilla, Associate Professor, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PID2020-114425RB
Record Dates: First submitted 2023-06-14; First posted 2023-09-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Emotion Regulation
Keywords: young adulthood; emotional Intelligence; well-being; Information and Communication Technologies (ICT)
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group (Experimental)
  Interventions: Behavioral: Participation in a socio-emotional competence program through a technological platform (EMOWELL)
- No Intervention: Control group (No Intervention)

INTERVENTIONS:
Behavioral: Participation in a socio-emotional competence program through a technological platform (EMOWELL) — (1) Participants who meet the inclusion criteria will be contacted. (2) Participants will answer the questionnaire battery (T1) (3) Participants will participate in the intervention by remotely playing the EMOWELL desktop serious game and the EMOWELL app. (4) They will answer the T2 questionnaires.
  Arms: Experimental: Intervention group

SUMMARY:
emoWELL is a serious game, that is, a video game designed to inform and train in skills and competencies in a more dynamic way. emoWELL focuses on understanding and developing healthy emotional regulation strategies to improve well-being.

DETAILED DESCRIPTION:
Computer-based videogame. The program has a graphic adventure format, where the player controls an avatar who embarks on a train journey. Throughout this journey, the train will make five different stops where the player will learn about emotional regulation through activities or puzzles, readings and different interventions with the game's characters. At the first stop, the player will receive psychoeducation about emotional regulation and the most frequent adaptive and maladaptive regulation strategies. In the next three areas, exercises will be carried out to apply these strategies on variables such as self-esteem, self-care, stress, time management and social support. Finally, in the last area, the player will review the different contents learned. In addition to the train and the five stops or areas described, the game includes the area of the avatar's house and a final scenario that will vary depending on the player's answers throughout the adventure, in order to highlight the most important learning and conclude the game. Therefore, emoWELL consists of 8 areas in total.

The intervention is carried out autonomously. In addition to the computer game, emoWELL is linked to a mobile application so that the user can practice, integrate and reinforce the knowledge learned in the remote game, being both platforms indispensable in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* To have signed the informed consent (or their legal tutors).
* Being between 18 and 29 years old.

Exclusion Criteria:

* Inability to understand the activities or the language used.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 385 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Inventory of the Dimensions of Emerging Adulthood (IDEA-S) | Time 1 (first month)
  The Spanish version is composed of 31 items. It is answered using a Likert scale from 1 (strongly disagree) to 3 (strongly agree). A higher score on a scale means a greater presence of these categories in the stage. It assesses the different characteristics of emerging adulthood: identity exploration, experimentation/possibilities, negativity/instability, other-centered, self-centered, feeling in between.
Inventory of the Dimensions of Emerging Adulthood (IDEA-S) | Time 2 (4th month)
  The Spanish version is composed of 31 items. It is answered using a Likert scale from 1 (strongly disagree) to 3 (strongly agree). A higher score on a scale means a greater presence of these categories in the stage. It assesses the different characteristics of emerging adulthood: identity exploration, experimentation/possibilities, negativity/instability, other-centered, self-centered, feeling in between.
Difficulties in Emotion Regulation Scale (DERS) | Time 1 (first month)
  The Spanish version is composed of 28 items. It is answered using a Likert scale from 1 (hardly ever) to 5 (almost always). This scale assesses difficulties associated of the emotion regulation process: emotional lack of control, life interference, lack of emotional attention, emotional confusion, and emotional rejection. Therefore, a higher score within each scale signals more difficulties in emotional regulation.
Difficulties in Emotion Regulation Scale (DERS) | Time 2 (4th month)
  The Spanish version is composed of 28 items. It is answered using a Likert scale from 1 (hardly ever) to 5 (almost always). This scale assesses difficulties associated of the emotion regulation process: emotional lack of control, life interference, lack of emotional attention, emotional confusion, and emotional rejection. Therefore, a higher score within each scale signals more difficulties in emotional regulation.
Emotion Regulation Questionnaire (ERQ) | Time 1 (first month)
  The scale is composed by 10 items. It is answered using a 7-point Likert scale.
Emotion Regulation Questionnaire (ERQ) | Time 2 (4th month)
  The scale is composed by 10 items. It is answered using a 7-point Likert scale.
Cognitive Emotion Regulation Questionnaire (CERQ-18) | Time 1 (first month)
  The instrument assesses cognitive strategies for emotional regulation. The version of the instrument used consists of 18 items and has five polytomous response options ranging from almost never (1) to always (5). The items are grouped into nine strategies: Rumination, Catastrophizing, Self-blaming, Blaming others, Putting in perspective, Acceptance, Positive focus, Positive reinterpretation, and Refocusing on plans; at a rate of two items per strategy.
Cognitive Emotion Regulation Questionnaire (CERQ-18) | Time 2 (4th month)
  The instrument assesses cognitive strategies for emotional regulation. The version of the instrument used consists of 18 items and has five polytomous response options ranging from almost never (1) to always (5). The items are grouped into nine strategies: Rumination, Catastrophizing, Self-blaming, Blaming others, Putting in perspective, Acceptance, Positive focus, Positive reinterpretation, and Refocusing on plans; at a rate of two items per strategy.
Psychological Well-Being Scales (PWBS) | Time 1 (first month)
  The Spanish version is composed of 29 items. It is answered using a Likert scale from 1 (totally agree) to 6 (totally disagree).
  A higher score on each scale indicates higher levels in the resulting dimensions of psychological well-being:
  Self-acceptance, Positive relationships, Autonomy, Environmental mastery, Purpose in life and Personal growth.
Psychological Well-Being Scales (PWBS) | Time 2 (4th month)
  The Spanish version is composed of 39 items. It is answered using a Likert scale from 1 (totally agree) to 6 (totally disagree).
  A higher score on each scale indicates higher levels in the resulting dimensions of psychological well-being:
  Self-acceptance, Positive relationships, Autonomy, Environmental mastery, Purpose in life and Personal growth.

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale (RSE) | Time 1 (first month)
  The RSE is an unidimensional instrument that consists of 10 items that assess self-esteem. Participants are asked to respond to each item using a four-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree." A higher score indicates higher levels of self-esteem.
Rosenberg Self-Esteem Scale (RSE) | Time 2 (4th month)
  The RSE is an unidimensional instrument that consists of 10 items that assess self-esteem. Participants are asked to respond to each item using a four-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree." A higher score indicates higher levels of self-esteem.
Brief Symptom Inventory (BSI-18) | Time 1 (first month)
  The instrument evaluates psychological distress, collected in three dimensions: anxiety, depression and somatization. It is composed of 18 items answered on a likert scale from 0 (Not at all) to 4 (Very much). Higher levels on each of these scales imply higher levels of anxiety, depression or somatization, respectively.
Brief Symptom Inventory (BSI-18) | Time 2 (4th month)
  The instrument evaluates psychological distress, collected in three dimensions: anxiety, depression and somatization. It is composed of 18 items answered on a likert scale from 0 (Not at all) to 4 (Very much). Higher levels on each of these scales imply higher levels of anxiety, depression or somatization, respectively.
Three-item loneliness scale (TILS) | Time 1 (first month)
  This scale evaluates the perception of loneliness. It is composed of three items answered on a Likert scale from 0 (Almost never) to 2 (Frequently). The higher the score, the greater the perception of loneliness.
Three-item loneliness scale (TILS) | Time 2 (4th month)
  This scale evaluates the perception of loneliness. It is composed of three items answered on a Likert scale from 0 (Almost never) to 2 (Frequently). The higher the score, the greater the perception of loneliness.
''Optimism questionnaire'' (COP) | Time 1 (first month)
  The last instrument presented is composed of 9 items. It evaluates the optimism of the participants. It is answered on a Likert scale from 1 to 5. A higher score implies higher levels of optimism.
''Optimism questionnaire'' (COP) | Time 2 (4th month)
  The last instrument presented is composed of 9 items. It evaluates the optimism of the participants. It is answered on a Likert scale from 1 to 5. A higher score implies higher levels of optimism.

CONTACTS AND LOCATIONS:
Locations (1):
- Spain, Valencia, Valencian Comunity, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Velert-Jimenez S, Sanchez-Sanchez H, Perez-Marin M, Gil-Gomez JA, Montoya-Castilla I. Emotion regulation intervention to promote well-being through a serious game (emoWELL): a study protocol for a randomised controlled trial in Spanish emerging adults. BMJ Open. 2025 Jul 16;15(7):e098230. doi: 10.1136/bmjopen-2024-098230. PMID 40669891